CLINICAL TRIAL: NCT00772551
Title: Evaluation of the Pharmacokinetics and Safety of Raltegravir and Ezetimibe When Co-administered to Male and Female Healthy Volunteers
Brief Title: Raltegravir and Ezetimibe PK Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Dr Marta Boffito, St Stephen's AIDS Trust
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SSAT027
Record Dates: First submitted 2008-10-10; First posted 2008-10-15 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: HIV
MeSH Terms: interventions — Raltegravir Potassium; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Raltegravir and ezetimibe
- 2 (Active Comparator)
  Interventions: Drug: Ezetimibe and raltegravir

INTERVENTIONS:
Drug: Raltegravir and ezetimibe — Group 1: raltegravir 400 mg orally twice daily for 10 days followed by 10 days of raltegravir 400 mg twice daily and ezetimibe 10 mg orally once daily for 10 days followed by a 10 days wash out period and ezetimibe 10 mg once daily for 10 days
  Arms: 1
Drug: Ezetimibe and raltegravir — Group2: ezetimibe 10 mg orally once daily for 10 days followed by ezetimibe 10 mg and raltegravir 400 mg orally twice daily for 10 days followed by a 10 days wash out period and raltegravir 400 mg twice daily for 10 days
  Arms: 2

SUMMARY:
Evaluation of the pharmacokinetics and safety of raltegravir and ezetimibe when co-administered to male and female healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
* Male or non-pregnant, non-lactating females
* Between 18 to 65 years, inclusive
* Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 1 month after the study

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
* Positive blood screen for hepatitis B and/or C antibodies
* Positive blood screen for HIV-1 and 2 antibodies
* Current or recent (within 3 months) gastrointestinal disease
* Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
* Exposure to any investigational drug or placebo within 4 weeks of first dose of study drug
* Consumption of grapefruit, or Seville oranges or any grapefruit or Seville orange containing product within one week of first dose of study drug and for the duration of the study
* Use of any other drugs, including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs.
* Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 30 days after the end of the treatment period
* Previous allergy to any of the constituents of the pharmaceuticals administered in this trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Steady state plasma concentrations of raltegravir and ezetimibe when given alone and in combination | 41 days

SECONDARY OUTCOMES:
Safety and tolerability of raltegravir and ezetimibe co-administration. Association between genetic polymorphisms in drug disposition genes and drug exposure. | 41 days

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- Chelsea and Westminster Hospital NHS Foundation Trust, London, London, United Kingdom